CLINICAL TRIAL: NCT06193200
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled Trial to Evaluate the Neurological Effects of EryDex on Subjects With Ataxia Telangiectasia (NEAT)
Brief Title: Evaluate the Neurological Effects of EryDex on Subjects With A-T
Acronym: NEAT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Quince Therapeutics S.p.A. (Industry)
Collaborators: Biotrial (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IEDAT-04-2022
Record Dates: First submitted 2023-12-11; First posted 2024-01-05 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Ataxia Telangiectasia
Keywords: Ataxia Telangiectasia; A-T; Louis-Bar syndrome; Cerebello-oculocutaneous telangiectasia
MeSH Terms: conditions — Ataxia Telangiectasia | interventions — dexamethasone 21-phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dexamethasone sodium phosphate (Experimental): IV infusion of dexamethasone sodium phosphate (DSP) encapsulated in autologous erythrocytes using the EryDex System (EDS)
  Interventions: Drug: Dexamethasone sodium phosphate
- Placebo (Placebo Comparator): IV infusion of placebo encapsulated in autologous erythrocytes using the EryDex System (EDS)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Dexamethasone sodium phosphate — Dexamethasone sodium phosphate encapsulated in autologous erythrocytes and administered via IV infusion
  Other Names: DSP
  Arms: Dexamethasone sodium phosphate
Other: Placebo — Placebo encapsulated in autologous erythrocytes and administered via IV infusion
  Arms: Placebo

SUMMARY:
This is an international, multi-center, randomized, prospective, double-blind, placebo-controlled, Phase 3 study, designed to assess the effect of EryDex (dexamethasone sodium phosphate [DSP] in autologous erythrocytes), administered by intravenous (IV) infusion once every 28 days, on neurological symptoms of patients with Ataxia Telangiectasia (A-T).

DETAILED DESCRIPTION:
The EryDex System (EDS) is a combination product that is used to load dexamethasone sodium phosphate (DSP) into autologous erythrocytes (EryDex) which is infused into the patient.

In the placebo arm, the subjects will receive autologous erythrocytes prepared with the EDS process using a placebo solution.

Upon completion of all screening assessments for eligibility, subjects meeting all selection criteria at baseline will be randomized in a 1:1 fashion to EryDex or placebo. Approximately 86 subjects 6- to 9-years-old, approximately 43 per group, will be randomized. Approximately 20 subjects 10 years of age and above, 10 per treatment group, may also be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of A-T
* In autonomous gait or is helped by periodic use of a support
* Genetic confirmation of A-T
* Body weight ≥15 kg

Exclusion Criteria:

* Participation in another clinical study
* Immune impairment
* History of severe impairment of the immunological system
* Current neoplastic disease or previous neoplastic disease not in remission for at least 2 years
* Severe or unstable pulmonary disease
* Uncontrolled diabetes
* Current chronic or acute significant renal and/or hepatic impairment
* Any previous oral or parenteral steroid use within 6 weeks before Baseline. Treatment with inhaled or intranasal steroids for asthma or allergies, as well as use of topical steroids will be permitted
* A disability that may prevent the subject from completing all study requirements

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2024-06-24 (Actual); Primary Completion 2025-12-17 (Actual); Study Completion 2025-12-17 (Actual)

PRIMARY OUTCOMES:
Rescored modified International Cooperative Ataxia Rating Scale (RmICARS) | Baseline to Visit 9 (approximately 6 months)
  Change of the RmICARS from baseline to Visit 9 compared to placebo (6 to 9 years old)

SECONDARY OUTCOMES:
Clinical Global Impression of Severity (CGI-S) | Baseline to Visit 9 (approximately 6 months)
  Change in CGI-S from baseline to Visit 9
Clinical Global Impression of Change (CGI-C) | Baseline to Visit 9 (approximately 6 months)
  Clinical Global Impression of Change (CGI-C) at Visit 9

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Thye, MD, Study Director — Quince Therapeutics S.p.A.
Locations (19):
- United States (4):
  - University of California Los Angeles (UCLA), Ataxia Center and HD Center of excellence, Los Angeles, California
  - The Johns Hopkins Hospital, Division of pediatric allergy and immunology, Baltimore, Maryland
  - Cincinnati Children's Hospital, Division of neurology, Cincinnati, Ohio
  - UT Health Houston, Department of pediatrics, division of child & adolescent neurology, Houston, Texas
- Copenhagen University Hospital, Rigshospitalet, Department of Pediatric Neurology, Copenhagen, Denmark
- Germany (2):
  - University Hospital Frankfurt, Pediatric and Adolescent Clinic, Frankfurt
  - IKF Pneumologie GmbH & Co. KG; Institut für klinische Forschung Pneumologie Clinical Research Center Respiratory Diseases, Frankfurt
- Italy (2):
  - Spedali Civili di Brescia, Pediatric immunology department, Brescia
  - Policlinico Umberto I, La sapienza University, Department of neurosciences and menthal health, Roma
- Oslo University Hospital, Rikshospitalet, Division of Pediatric and Adolescent Medicine, Norwegian National Unit for Newborn Screening, Oslo, Norway
- Poland (2):
  - MedPolonia sp zoo, Poznan
  - Instytut "Pomnik-Centrum Zdrowia Dziecka", Immunology clinic, Warsaw
- Spain (2):
  - Hospital Universitari Vall d'Hebron, Department of pediatric neurology, Barcelona
  - Hospital Universitario La Paz, Department of pediatric neurology, Madrid
- University Children's Hospital Zürich - Eleonore Foundation, Zurich, Switzerland
- United Kingdom (4):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - St George's University Hospitals NHS Foundation Trust, Centre for Neonatal and Paediatric Infection, London
  - Great Ormond Street Hospital for Children, Zayed Centre for Research, London
  - Nottingham Children's Hospital, Queen's Medical Center, Children's neurology, Nottingham

IPD SHARING:
Plan to Share IPD: No